CLINICAL TRIAL: NCT04427683
Title: Effects of a Brief Mindful Parenting Program for Hong Kong Chinese Impacted by Social Unrest: A Randomised Trial
Brief Title: Effects of a Brief Mindful Parenting Program for Hong Kong Chinese Impacted by Social Unrest
Acronym: MPHKC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SR2020.A6.004
Record Dates: First submitted 2020-06-05; First posted 2020-06-11 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2020-06

CONDITIONS: Mental Health Issue
Keywords: parent depression; parent mental health; mindfulness-based intervention

STUDY DESIGN:
Intervention Model Description: Recruited and eligible participants will be randomised into an intervention group and a wait-list control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief mindful parenting program (Experimental): The program will consist of a four-session and last for eight hours integrating mindfulness skills and psychoeducation in managing stress under social unrest and promoting strategies for emotion regulation, conflict management, and self-care.
  Interventions: Behavioral: Brief mindful parenting program
- Wait-list control group (Other): A four-minute educational video will be distributed to the participants who accept the randomisation. It includes brief information on mental health. After the participants from experimental group complete the intervention, those in wait-list control group will receive the same intervention.
  Interventions: Behavioral: Brief mindful parenting program

INTERVENTIONS:
Behavioral: Brief mindful parenting program — Mindfulness exercise include formal and informal mindfulness exercises, and additional exercise for coping with anger and arousing emotions. Psychoeducation includes understanding relationship between thoughts and feelings, fight or flight responses and adaptive coping in parenting relationship.

SUMMARY:
A four session mindful parenting workshop is designed to promote parental mental health during the social unrest in 2020. This study is conducted to investigate the outcome of the program. It is a randomised control trial design and will be conducted in five sites in Hong Kong. An estimated 340 parents will be recruited and randomised into an intervention group and a wait-list control group. The primary outcome is parental depression. Secondary outcomes include parental anxiety and post-traumatic stress, negative emotions, family functioning, family conflict and mindful parenting. Exposure to social unrest will be measured and the relationship to mental health and effects of the program will be examined.

DETAILED DESCRIPTION:
Design: With a self-administered screening for depression (PHQ-9), parents with a subclinical cutoff score or above will be eligible to participate in a four-session parent workshop. The same program will be provided in five locations in Hong Kong. A waitlist-control randomised controlled trial will be used to evaluate the outcomes of the program. An estimated 340 parents will be recruited and randomised into an intervention group and a wait-list control group. The sample estimation is based on an expected effect size of .33 for family functioning in the PI's pilot study, with an estimated drop-out rate of 15%, a two-tailed α error of 5%, 80% power, and a test of two independent groups.

Measures: (1) Exposure to social unrest will be measured using the Political Life Events Scale. The scale contains 20 items related to stressful events, to which respondents report exposure by answering yes or no. In view of the local context, only 16 items will be used. (2) Negative emotions about social unrest will be measured by the three items developed by Halperin et al. The items assess the intensity of negative emotions (hatred, anger, despair) in the context of social unrest, with responses given on a Likert-type scale ranging from 1 (not at all) to 10 (very strong). (3) Depression and anxiety symptoms will be assessed by the Patient Health Questionnaire (PHQ-9) and the Generalized Anxiety Disorder 7-item (GAD-7) scale. (4) Traumatic stress will be assessed by the International Trauma Questionnaire (ITQ), a 6-item self-report measure of the major symptoms of post-traumatic stress. The ITQ has been translated into Chinese and validated for screening of post-traumatic stress. (5) Family functioning will be assessed by the Family APGAR (Adaptation, Partnership, Growth, Affection, Resolve) scale (APGAR). The 5-item scales uses a 3-point response scale (0 = hardly ever and 2 = almost always). A cutoff for severe family dysfunction is available for Chinese families. (6) Family conflict will be measured by the Conflict Tactics Scale (CTS-2), a self-report measure of behavioural assault or psychological aggression among family members. It has been used in studies of conflict between adolescents and parents.

ELIGIBILITY:
Inclusion Criteria:

* parents of adolescents at aged between 10 to 21
* a score of PHQ-9 of 2 or above

Exclusion Criteria:

* parents with self-reported psychosis, alcohol or substance abuse, individual or family crisis in last six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Depression | Change from pre-intervention (T0), to 1-month follow up (T1), and to 3-month follow-up (T2).
  Self-administered measure Patient Health Questionnaire (PHQ-9), 9 items, sum of scores range from 0 to 27, the higher the score, the more severe in depressive symptoms

SECONDARY OUTCOMES:
Anxiety | Change from pre-intervention (T0), to 1-month follow up (T1), and to 3-month follow-up (T2).
  Self-administered measure Generalized Anxiety Disorder 7-item scale (GAD-7), 7 items, sum of scores from 0 to 21, the higher the score, the more severe in the anxiety symptoms
Post-traumatic stress | Change from pre-intervention (T0), to 1-month follow up (T1), and to 3-month follow-up (T2).
  self-administered measure International Trauma Questionnaire (ITQ), 6 items, sum of scores range from 0 to 24, the higher the score, the more severe the post-traumatic stress symptoms
family functioning | Change from pre-intervention (T0), to 1-month follow up (T1), and to 3-month follow-up (T2).
  self-administered measure Family APGAR (Adaptation, Partnership, Growth, Affection, Resolve) scale (APGAR), 5 items, sum of the scores range from 0 to 10, the higher the score, the better in family functioning
family conflict | Change from pre-intervention (T0), to 1-month follow up (T1), and to 3-month follow-up (T2).
  self-administered measure Conflict Tactics Scale (CTS-2), 16 items, sum of scores range from 0 to 112, the higher the score, the more stronger intensity the family conflict is
mindful parenting | Change from pre-intervention (T0), to 1-month follow up (T1), and to 3-month follow-up (T2).
  self administered measure, Interpersonal Mindfulness in Parenting scale, 6 items in nonjudgmental acceptance in parenting and 4 items in listening with full attention, sum of scores range from 6 to 30 for nonjudgmental acceptance in parenting, and 6 to 20 for listening with full attention, the higher the score, the stronger the interpersonal mindfulness level is

CONTACTS AND LOCATIONS:
Overall Officials: Herman, Hay-ming LO, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- LO, Herman Hay-ming, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The protocol will be published in an open access academic journal.

REFERENCES:
- [Derived] Lo HHM, Lau ENS, Tam CHL, Ngai SW, Chan SHW, Leung BFH, Wong ET, Wong EWY, Wong GOC, Cho WC, Tsang AWK, Singh NN. Effects of a Mindful Parenting Workshop for Parents of Adolescents and Young Adults Following Social Unrest in Hong Kong. Mindfulness (N Y). 2022;13(1):248-261. doi: 10.1007/s12671-021-01790-7. Epub 2021 Dec 2. PMID 34873419

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-28): https://cdn.clinicaltrials.gov/large-docs/83/NCT04427683/Prot_SAP_001.pdf
  • Informed Consent Form (2019-11-28): https://cdn.clinicaltrials.gov/large-docs/83/NCT04427683/ICF_000.pdf